CLINICAL TRIAL: NCT06259344
Title: Effect of Pain Science Education Administered in Full or Fractioned Dosage Modes Associated With Conventional Treatment on Pain Intensity and Disability for Temporomandibular Disorders: a Randomized Controlled Trial
Brief Title: Pain Science Education Administered in Full or Fractioned Dosage Modes for Temporomandibular Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Thais Chaves, Ph.D, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77273924.9.0000.5504
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Experimental: Fractioned Pain Science Education (PSE) program + Manual Therapy + Orofacial and Neck Motor Exercises (ONE) (FPSE) Six sessions of 15 minutes each of a workshop on PSE will be administered. Two protocols of ONE and Manual Therapy (MT) and ONE will be administered. The exercises will be administered for six weeks, twice a week. Half of the sessions will include orofacial therapy and exercises and half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
  Active Comparator: Full Dosage Mode PSE (FDPSE) + MT + ONE Two sessions of 45 minutes (90 minutes) of PSE will be administered. Two protocols of ONE and MT will be administered. The exercises will be administered for six weeks, twice a week. Half of the sessions will include orofacial therapy and exercises and half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractioned Pain Science Education + Manual Therapy + Orofacial and Neck Exercises (Active Comparator): All participants in this arm will initially receive six sessions in which a workshop on PSE will be administered and discussed. A power-point presentation with metaphors and animated videos will be employed. The PSE program will be held in 6 sessions of 15 minutes each. Two protocols of Orofacial Exercises and Manual Therapy and of Neck Motor Control will be adopted in the present study. The exercises will be administered during six weeks, twice a week. One session will run in the outpatient clinic and the other will be home based. Half of the sessions will consist of orofacial therapy and exercises and the other half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
  Interventions: Behavioral: Fractioned Pain Science Education (FPSE); Other: Manual Therapy; Other: Orofacial and Neck Exercises (ONE)
- Full Dosage Pain Science Education + Manual Therapy + Orofacial and Neck Exercises (Experimental): All participants in this arm will initially receive two sessions in which a workshop on PSE will be administered and discussed. A power-point presentation with metaphors and animated videos will be employed. The PSE program will be held in 2 sessions of 45 minutes each one. Two protocols of Orofacial Exercises and Manual Therapy and of Neck Motor Control will be adopted in the present study. The exercises will be administered during six weeks, twice a week. One session will run in the outpatient clinic and the other will be home based. Half of the sessions will consist of orofacial therapy and exercises and the other half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
  Interventions: Behavioral: Full Dosage Mode Pain Science Education (FDPSE); Other: Manual Therapy; Other: Orofacial and Neck Exercises (ONE)

INTERVENTIONS:
Behavioral: Fractioned Pain Science Education (FPSE) — Pain Science Education (PSE) will be administered in workshop sessions with interactive presentations, using different resources as metaphors and videos. It will be held in 2 sessions of 45 minutes each, covering 6 topics of Explain Pain and Explain Pain Supercharged books.
  Arms: Fractioned Pain Science Education + Manual Therapy + Orofacial and Neck Exercises
Behavioral: Full Dosage Mode Pain Science Education (FDPSE) — Pain Science Education (PSE) will be administered in workshop sessions with interactive presentations, using different resources as metaphors and videos. It will be held in 6 sessions of 15 minutes each, covering 6 topics of Explain Pain and Explain Pain Supercharged books.
  Arms: Full Dosage Pain Science Education + Manual Therapy + Orofacial and Neck Exercises
Other: Manual Therapy — Intraoral temporalis release, Intraoral medial and lateral pterygoid (origin) technique and Intraoral sphenopalatine ganglion technique.
Other: Orofacial and Neck Exercises (ONE) — Orofacial Exercises: Mandibular body-condylar cross-pressure chewing technique; Post-isometric relaxation stretches-laterotrusion and opening (10 times/session; 10 seconds).
  Neck Motor Control Exercises: Bracing exercises (6 hierarchical levels - HL). Extreme range of motion exercises (stable spine). Cervical isometric exercises (5 HL) directly forward, obliquely, toward right and left, and directly backward (stable spine - elastic resistive bands). Functional training with elastic resistance and exercise balls on unstable surfaces (8 HJ). The progress in each exercise domain will happen when sustaining the contraction for 10 seconds, 10 times.

SUMMARY:
Temporomandibular Disorders (TMD) are a collection of musculoskeletal disorders which affect the masticatory structures and have a multifactorial etiology. A biopsychosocial approach is recommended for the management of these disorders including different interventions like exercise, manual therapy and pain education. The aim of this study is to compare the effect of a full dosage mode pain science education program (2 initial sessions of 45 minutes) versus a fractioned dosage format (6 sessions of 15 minutes) combined with manual therapy and orofacial exercises on primary outcomes - pain intensity and disability - and secondary outcomes - mandibular range of motion, pain-related self-efficacy, kinesiophobia, global perception of improvement, empathy, knowledge about pain neuroscience, beliefs about pain, exercise adherence, and catastrophizing - in patients with chronic painful TMD. This study will be a randomized controlled trial with a sample of 148 participants. Individuals will undergo a screening process to identify those with TMD diagnosis according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD), aged 20 to 60 years, of both genders, and then the volunteers will be randomized into two groups (G1: Full dosage mode pain science education program + Manual therapy/orofacial and neck motor exercises vs. G2: Fractioned dosage mode pain science education program + Manual therapy/orofacial and neck motor exercises). These volunteers will be recruited in the city of São Carlos, SP. The intervention will take place twice a week for 8 weeks, administered by a single therapist, each session lasting 1 hour. The primary outcomes will be pain intensity and disability, assessed using the numerical pain rating scale and the Craniofacial Pain and Disability Inventory (CFP-DI), respectively, and the secondary outcomes will be mandibular range of motion, pain-related self-efficacy, kinesiophobia, global perception of improvement, empathy, knowledge about pain neuroscience, beliefs about pain, exercise adherence, and catastrophizing, assessed using the Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD), Global Perceived Effect of Improvement scale, Pain Self-Efficacy Questionnaire (PSEQ), CARE Empathy Scale, and Pain Catastrophizing Scale (PCS). For statistical analysis, a Generalized Estimated Equations considering time and groups as factors will be used. A significance level of p<0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 60 years;
* painful TMD (confirmed by applying DC/TMD);
* complaint of pain with a minimum intensity of 3 (on a scale of 0 to 10) present for at least 3 months;
* fluency to speak and understand Brazilian Portuguese (Mini Cog instrument to assess cognitive capacity and the Cloze Test to certify textual reading comprehension)

Exclusion Criteria:

* history of tumors in the orofacial region;
* central and peripheral neurological diseases;
* uncontrolled psychiatric illnesses;
* pregnant women;
* presence of toothache, neuralgia or chronic painful conditions in the head region, orofacial region or systemic pain (for example, fibromyalgia, osteoarthritis, osteoarthritis or rheumatological diseases);
* report of previous major surgeries in the craniofacial region, such as orthognathic surgeries, TMJ surgeries, or resulting from post-trauma corrections;
* history of major trauma involving the cervical or craniofacial region (facial trauma, whiplash injuries, etc.);
* individuals undergoing physiotherapeutic treatment up to 6 months before the start of this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-12-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity | Immediately after treatment, three-, six- and twelve- month follow-up
  The Numerical Pain Rating Scale will be used to assess pain intensity in this trial. It consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change in Orofacial Pain related Disability | Immediately after treatment, three-, six- and twelve- month follow-up
  The Craniofacial Pain and Disability Inventory (CF-PDI) is a self-administered questionnaire that measures the outcomes of pain and disability related to craniofacial pain. It demonstrated a good structure, internal consistency, reproducibility, and construct validity. Also, the Brazilian Portuguese version showed acceptable psychometric measurements. It consists of 21 items, with a score ranging from 0 to 63 points. Each question is scored on a 4-point ordinal scale, ranging from 0 to 3. A higher score reflects higher disability levels.

SECONDARY OUTCOMES:
Change in Pain-Related Self-efficacy | Immediately after treatment, three-, six- and twelve- month follow-up
  The Pain Self-Efficacy Questionnaire (PSEQ) will be used to measure pain self-efficacy beliefs (ability to function despite pain). Each item is rated by selecting a number on a 7-point scale, where 0 equals ''not at all confident'' and 6 equals ''completely confident''. A total score is calculated by summing the scores for each of the 10 items, resulting in a maximum possible score of 60. Higher scores reflect stronger self-efficacy beliefs. In the study analyzing the measurement properties of the Brazilian Portuguese version, the reliability of the PSEQ was considered adequate (the correlation divided in half was 0.76 and the internal consistency was 0.90).
Change in Kinesiophobia | Immediately after treatment, three-, six- and twelve- month follow-up
  The kinesiophobia outcome will be measured using the Tampa Scale For Kinesiophobia for Temporomandibular Disorders (TSK/TMD-Br). This is an 18-item self-report instrument that assesses fear of movement. The version translated into Brazilian Portuguese, TSK/TMD-Br, has 12 items. Each item is scored on a 4-point Likert scale, ranging from "strongly disagree" (score = 1) to "strongly agree" (score = 4). Responses are summed to produce a total score in which higher values reflect greater fear of movement (12-48 points) The TSK/TMD has good reliability (CCI = 0.66-0.83) and acceptable validity values (VISSCHER et al., 2010). Internal consistency analysis demonstrated adequate Cronbach's α values (>0.70) for all domains and reliability demonstrated excellent ICC values for all domains (ICC>0.75).
Change in Global Perceived Effect of Improvement | Immediately after treatment, three-, six- and twelve- month follow-up
  The Global Perceived of Effect of improvement has 11 points and ranges from -5 ("much worse") to 0 ("no change") to +5 ("completely recovered"). A higher score indicates greater recovery from the condition.
Status of Empathy with the care provider | Immediately after treatment
  The CARE Empathy Scale measures the degree of perception of empathy on the part of the patient, which can influence the effectiveness of the intervention. The instrument consists of 10 items, with additional explanations of colloquial language, aiming to facilitate understanding of the questions. The answers range from 1 "poor" to 5 "excellent". All item values are then added together, providing a final score between 10 and 50. The version translated into Brazilian Portuguese has a Cronbach's alpha coefficient of 0.867.
Previous and acquired knowledge about pain neuroscience | Immediately after treatment, three-, six- and twelve- month follow-up
  The Neurophysiology of Pain Questionnaire (NPQ) will be used to verify learning related to the pain neuroscience education program. The 19 items have the following response options: true, false, undecided. Each correct question receives a score of 1. Incorrect answers and/or answers marked as undecided are not scored. The NPQ is scored out of 19 with 1 point awarded for each correct response. A score of 0 is attributed to incorrect responses and those marked as undecided. The internal consistency analysis revealed a reliability value of alpha = 0.63.
Beliefs about pain | Immediately after treatment, three-, six- and twelve- month follow-up
  The Concept Of Pain Inventory for Adults (COPI-ADULT) will be administered to assess participants' beliefs about pain. This instrument consists of 13 items. The items are presented on a 5-point Likert scale: 0 strongly disagree; 1 disagree; 2 I'm not sure; 3 agree and 4 strongly agree. Higher COPI-Adult scores reflect greater alignment with contemporary pain science (total scores can range from 0 to 52). It presents acceptable internal consistency (α=0.78) and good test-retest reliability at 1 week (intraclass correlation coefficient of 0.84 (95% confidence interval: 0.71-0.91).
Previous and current exercise adherence behaviour | Immediately after treatment, three-, six- and twelve- month follow-up
  The Exercise Adherence Assessment Scale (EARS-Br) is made up of six items that assess the exercise behavior adherence and has 5 possible answer options (0 = completely agree to 4 = completely disagree), the total score ranges from 0 to 24 points, the higher the score, the greater the adherence. The structure of the single-factor EARS-Br instrument with 6 items showed acceptable fit indices (comparative fit index and goodness-of-fit index > 0.90 and root mean square error of approximation < 0.08). The EARS-Br scale showed acceptable internal consistency (α = 0.88) and excellent reliability (ICC = 0.91). A Minimally Important Change (MIC) of 5.5 in the EARS-Br total score was considered a significant change in adherence behavior (AUC = 0.82). Moderate accuracy (AUC = 0.89) was obtained for a total EARS cutoff score of 17/24 after home exercise prescription. Sensitivity and specificity are also acceptable (greater than 80%).

CONTACTS AND LOCATIONS:
Overall Officials: Thais Chaves, Ph.D, Study Chair — Federal University of São Carlos - UFSCar
Locations (1):
- Federal University of São Carlos - Department of Physical Therapy, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguiar ADS, Moseley GL, Bataglion C, Azevedo B, Chaves TC. Education-Enhanced Conventional Care versus Conventional Care Alone for Temporomandibular Disorders: A Randomized Controlled Trial. J Pain. 2023 Feb;24(2):251-263. doi: 10.1016/j.jpain.2022.09.012. Epub 2022 Oct 8. PMID 36220481
- [Background] Calixtre LB, Moreira RF, Franchini GH, Alburquerque-Sendin F, Oliveira AB. Manual therapy for the management of pain and limited range of motion in subjects with signs and symptoms of temporomandibular disorder: a systematic review of randomised controlled trials. J Oral Rehabil. 2015 Nov;42(11):847-61. doi: 10.1111/joor.12321. Epub 2015 Jun 7. PMID 26059857
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Herrera-Valencia A, Ruiz-Munoz M, Martin-Martin J, Cuesta-Vargas A, Gonzalez-Sanchez M. Effcacy of Manual Therapy in TemporomandibularJoint Disorders and Its Medium-and Long-TermEffects on Pain and Maximum Mouth Opening:A Systematic Review and Meta-Analysis. J Clin Med. 2020 Oct 23;9(11):3404. doi: 10.3390/jcm9113404. PMID 33114236
- [Background] Leake HB, Mardon A, Stanton TR, Harvie DS, Butler DS, Karran EL, Wilson D, Booth J, Barker T, Wood P, Fried K, Hayes C, Taylor L, Macoun M, Simister A, Moseley GL, Berryman C. Key Learning Statements for Persistent Pain Education: An Iterative Analysis of Consumer, Clinician and Researcher Perspectives and Development of Public Messaging. J Pain. 2022 Nov;23(11):1989-2001. doi: 10.1016/j.jpain.2022.07.008. Epub 2022 Aug 4. PMID 35934276
- [Background] Maixner W, Diatchenko L, Dubner R, Fillingim RB, Greenspan JD, Knott C, Ohrbach R, Weir B, Slade GD. Orofacial pain prospective evaluation and risk assessment study--the OPPERA study. J Pain. 2011 Nov;12(11 Suppl):T4-11.e1-2. doi: 10.1016/j.jpain.2011.08.002. No abstract available. PMID 22074751
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Romm MJ, Ahn S, Fiebert I, Cahalin LP. A Meta-Analysis of Therapeutic Pain Neuroscience Education, Using Dosage and Treatment Format as Moderator Variables. Pain Pract. 2021 Mar;21(3):366-380. doi: 10.1111/papr.12962. Epub 2020 Nov 22. PMID 33131210
- [Background] Salazar-Mendez J, Nunez-Cortes R, Suso-Marti L, Ribeiro IL, Garrido-Castillo M, Gacitua J, Mendez-Rebolledo G, Cruz-Montecinos C, Lopez-Bueno R, Calatayud J. Dosage matters: Uncovering the optimal duration of pain neuroscience education to improve psychosocial variables in chronic musculoskeletal pain. A systematic review and meta-analysis with moderator analysis. Neurosci Biobehav Rev. 2023 Oct;153:105328. doi: 10.1016/j.neubiorev.2023.105328. Epub 2023 Jul 27. PMID 37516218
- [Background] Slade GD, Ohrbach R, Greenspan JD, Fillingim RB, Bair E, Sanders AE, Dubner R, Diatchenko L, Meloto CB, Smith S, Maixner W. Painful Temporomandibular Disorder: Decade of Discovery from OPPERA Studies. J Dent Res. 2016 Sep;95(10):1084-92. doi: 10.1177/0022034516653743. Epub 2016 Jun 23. PMID 27339423
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Derived] Spavieri JHP, de Lima TC, Pereira RBR, Chaves TC. Effect of pain science education administered condensed or longitudinally associated with manual therapy and exercises on pain intensity and disability for Temporomandibular Disorders: a randomized controlled trial. Trials. 2025 Dec 18. doi: 10.1186/s13063-025-09320-9. Online ahead of print. PMID 41413604